CLINICAL TRIAL: NCT06228508
Title: Molecular Diagnosis of Lung Cancer Via Bronchoscopy: The Significance of Bronchial Liquid Biopsy (ctDNA and ctRNA)
Acronym: BiliBro
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231133
Record Dates: First submitted 2023-11-06; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Bronchial ctDNA; Bronchial ctRNA; Bonrchoscopy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ctDNA and ctRNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The management of lung cancer is a major public health challenge. Molecular anomaly testing is recommended from the early stages for optimal and personalized care of all lung adenocarcinomas and non-smoker lung cancers. The search for these anomalies relies on increasingly advanced and sensitive analysis techniques, particularly Next-Generation Sequencing (NGS), which can simultaneously detect various molecular abnormalities in both DNA and RNA, including point mutations, complex mutations, rearrangements, and amplifications. These techniques are predominantly performed on biopsy specimens embedded in paraffin. However, these biopsies may require invasive and sometimes iatrogenic procedures, and their feasibility, quantity, and quality of the samples can be limited. The turnaround time for analysis results from the time of biopsy is typically around 2 to 3 weeks.

In recent years, alongside the improvement in the sensitivity of molecular analysis techniques, liquid biopsy has emerged as a valuable approach, particularly in the analysis of circulating tumor DNA (ctDNA). ctDNA is a non-invasive diagnostic biomarker that has been validated for detecting targetable molecular anomalies similar to those detected by "conventional" biopsies. ctDNA can be detected in plasma through a simple blood draw, as well as in cerebrospinal fluid, urine, saliva, or any other "liquid" sample from the patient. The concordance between mutations identified in the tumor and those detected in the blood exceeds 90% specificity in numerous studies. However, the sensitivity of ctDNA detection varies depending on the stage of the disease and the sensitivity of the detection technique used.

The utility of bronchial ctDNA is currently underexplored. However, there is a rationale for investigating ctDNA as close as possible to the cancerous lesion at the bronchial level. Bronchial ctDNA could play a role in molecular diagnosis for distal lesions not visible through endoscopy and could also help reduce costs and turnaround time for molecular diagnosis in larger tumors.

The objective of this study is to evaluate the utility of liquid biopsy (ctDNA and ctRNA) during bronchoscopy in the molecular diagnosis and management of bronchial carcinomas. This is a prospective multicenter French study that will include 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients Referred for Bronchoscopy at TNN or PSL for Diagnostic Evaluation or Follow-up of Known or Suspected Lung Cancer.
* Age >18 years.
* Informed, Written, and Signed Consent.
* Participants must be covered by a national health insurance scheme.

Exclusion Criteria:

* Patient Refusal
* Patient benefiting from legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Undergoing Bronchoscopy for Diagnostic Evaluation or Follow-up of Lung Cancer
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Sensibility of bronchial ctDNA | Through study completion, an average of 6 month
  Calculation of the sensitivity of bronchial ctDNA for the molecular diagnosis of lung cancers

SECONDARY OUTCOMES:
Diagnostic Performance of ctDNA Molecular Testing | Through study completion, an average of 6 month
  Specificity; Positive Predictive Value; Negatice Predictive Value
Diagnostic Performance of ctDNA Molecular Testing | Through study completion, an average of 6 month
  Sensibility; Specificity; Positive Predictive Value; Negatice Predictive Value
Comparing Turnaround Time of Molecular Biology Results | Through study completion
  Time of Molecular Biology Results for Bronchial ctDNA and ctRNA (versus Standard Histology)
Comparison of Performance between Bronchial ctDNA and Blood ctDNA when Available | Through study completion, an average of 6 month
  Calculation of the concordance rate between these 2 methods.
Evaluating Analysis Modalities in Liquid Biopsy Techniques | Through study completion, an average of 6 month
  Description of the methods of the analysis technique using the supernatant vs pellet
Subgroup Analysis of Diagnostic Performance of Bronchial ctDNA and ctRNA | Through study completion, an average of 6 month
  Description of the mutations found in the lung cancers

CONTACTS AND LOCATIONS:
Overall Officials: Vincent FALLET, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Pneumologie et Oncologie Thoracique - Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided